CLINICAL TRIAL: NCT02957526
Title: Use of an Innovative Mobile Health Application to Improve Health Outcomes for Breast Cancer Patients
Brief Title: Web-Base App To Improve Aromatase Inhibitor Adherence
Acronym: AETAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: University of Tennessee West Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-04088-XP
Record Dates: First submitted 2016-10-31; First posted 2016-11-07 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2016-10

CONDITIONS: Breast Neoplasm Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- App (Experimental): The web-based app will be used to ask participants about their aromatase inhibitor use in the previous 7 days and ask about treatment-related adverse symptoms, or changes in the severity of symptoms. Participants will receive reminders via text or email to use the app once per week. All participants will be followed for a 6-8 weeks (depending on the data of participants' in-clinic follow-up visit) and will be asked to complete a baseline survey at enrollment and a follow-up survey at their 6-8 week in-clinic follow-up visit.
  Interventions: Behavioral: Prompts to report symptoms via study app; Behavioral: Clinical Alerts
- Usual Care (Active Comparator): Participants will have access to the web-based app, but will not receive reminders. All participants will be followed for a 6-8 weeks (depending on the data of participants' in-clinic follow-up visit) and will be asked to complete a baseline survey at enrollment and a follow-up survey at their 6-8 week in-clinic follow-up visit.
  Interventions: Behavioral: Clinical Alerts

INTERVENTIONS:
Behavioral: Prompts to report symptoms via study app — Weekly prompts to report aromatase inhibitor use in the previous 7 days and treatment-related adverse symptoms via the web-enabled study app.
  Arms: App
Behavioral: Clinical Alerts — : Reported symptoms may trigger an email alert to the participant's care team based on predetermined thresholds. Alerts based on certain response thresholds are generated to inform the patient's care team of any concerning responses or trends that emerge from the patient reported outcomes. These alerts will inform providers of particular patient-related adverse events or symptoms requiring an intervention prior to the point that emergent medical care is needed. Information in the alert emails will include the participant's Medical Reference Number (MRN), initials, date of birth, and details about the symptom(s) that generated the alert. Pod nurses instructed to respond to any clinical alerts (sent via email) as soon as possible following standard of care.

SUMMARY:
The purpose of this study will be to test the use of a web-based mobile application (app) initiated at the time of the initial prescription to an aromatase inhibitor to improve communication and management of treatment-related adverse symptoms among patients with hormone-receptor positive breast cancer.

DETAILED DESCRIPTION:
About 1 in 8 women are diagnosed with breast cancer during their lifetime; among them over 80% have hormone receptor-positive (HR+) tumors. Long-term aromatase inhibitors are commonly prescribed to women with HR+ breast cancer after surgery, chemotherapy, and/or radiation to lower cancer recurrence rates and improve survival. Despite the potential improvement in survival outcomes, recent evidence suggests that aromatase inhibitor adherence and persistence rates are low. Multiple studies point to adverse side effects of adjuvant therapies as a key reason for lower adherence or premature discontinuation. Patients who do not take the full amount of their medication as prescribed or who discontinue their aromatase inhibitor treatment early do not receive the full intended treatment benefits, and consequently are at increased risk for all-cause mortality, cancer death, and recurrence. Monitoring of adverse effects and symptoms, especially between clinic visits, could help healthcare providers better manage symptoms and increase long-term treatment adherence. Evidence indicates that patients generally experience most adverse effects early in their treatment, typically within the first six months. We plan to enroll 20 subjects per study arm, for a total of 40 participants. Potential subjects for recruitment will be identified from the electronic health records system of the West Cancer Center. Physicians and nurses at the West Cancer Center refer potentially eligible patients to the study nurse coordinator. The nurse will review eligibility criteria with patients and provide an overview of the research study and seek informed consent. Patients who provide informed consent will immediately be asked to complete a brief baseline survey about their preferences for receiving prompts, either via email or via cell phone using a text message. After survey administration, all patients will be registered in the mobile health app, which will be used report medication adherence and any related adverse symptoms. Study participants will be randomized into one of two arms: 1) active prompts to use the study app or 2) use of study app, but no prompts. All participants will be followed for a minimum of 6-8 weeks (depending on their scheduled follow-up visits at the center) and will be asked to complete a follow-up survey during or shortly after their scheduled in-clinic appointment at the end of the study. Baseline and follow-up questionnaires will collect data on quality of life (FACT-ES), health literacy, and demographics. The web-based app will be used to ask patients about medication adherence in the previous 7 days, any new symptoms, or changes in the severity of symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients (age≥18)
2. Diagnosed with early stage (I-III) HR+ breast cancer
3. New prescription for an aromatase inhibitor
4. Have a mobile device with a data plan or a home computer with Internet
5. Have a valid email address
6. Willing to complete brief weekly symptom reports on the app

Exclusion Criteria:

1. Unable to communicate in English
2. Patients with prior use of adjuvant endocrine therapy will also be excluded
3. Patients concurrently undergoing surgery, chemotherapy or radiation will also be excluded
4. Current diagnosis of rheumatoid arthritis
5. Chronic daily narcotic usage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Aromatase inhibitor adherence using the four-item Morisky Medication Adherence Scale | 6-8 weeks
  The primary data analysis will adhere to the intention-to-treat principle and in the final analysis, the participants will be categorized according to their initial randomization. Investigators will measure differences in aromatase inhibitor adherence at end of the study between the two study arms using the four-item Morisky Medication Adherence Scale.
Aromatase inhibitor adherence using the single item MAR-Scale global question | 6-8 weeks
  The primary data analysis will adhere to the intention-to-treat principle and in the final analysis, the participants will be categorized according to their initial randomization. Investigators will measure differences in aromatase inhibitor adherence at end of the study between the two study arms using the Medication Reasons Adherence (MAR-Scale) single item global question which asks about medication adherence in the past 7 days.

SECONDARY OUTCOMES:
Symptom Burden | 6-8 weeks
  Investigators also plan to carry out a secondary analysis, which will adhere to the intention-to-treat principle and in the final analysis, the participants will be categorized according to their initial randomization. Investigators will measure relative changes in adverse symptom burden (measured using surveys collected at baseline and at follow-up 6-8 weeks after the intervention using the FACT-ES questionnaire) between the two study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Graetz, PhD, Principal Investigator — University of Tennessee
Locations (2):
- United States (2):
  - West Cancer Center, MIDTOWN, 1588 Union Ave., Memphis, Tennessee
  - West Cancer Center, EAST MEMPHIS, 7945 Wolf River Blvd, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Graetz I, McKillop CN, Stepanski E, Vidal GA, Anderson JN, Schwartzberg LS. Use of a web-based app to improve breast cancer symptom management and adherence for aromatase inhibitors: a randomized controlled feasibility trial. J Cancer Surviv. 2018 Aug;12(4):431-440. doi: 10.1007/s11764-018-0682-z. Epub 2018 Feb 28. PMID 29492753